CLINICAL TRIAL: NCT04286789
Title: A Randomized, Double-blind, Parallel, Vehicle Controlled, Repeat Dose Comparative Phase 1b Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ORTD-1 in Rheumatoid Arthritis Patients With Mild Disease Managed With DMARDs
Brief Title: Randomized, Double-blind, Vehicle Controlled, Repeat Dose Comparative Study in RA Patients Managed With DMARDs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oryn Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ORTD1-002
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rhesus-theta-defensin-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ORTD-1-Low Dose (Experimental): 5.6 mg/0.45 mL of active study drug
  Interventions: Drug: Low dose ORTD-1
- Vehicle Control -Low Dose (Placebo Comparator): Vehicle (Identical formulation without the active DP)
  Interventions: Drug: Low dose vehicle control
- ORTD 1-High Dose (Experimental): 22.5 mg/1.8 mL of active study drug
  Interventions: Drug: High dose ORTD-1
- Vehicle Control -High Dose (Placebo Comparator): Vehicle (Identical formulation without the active DP)
  Interventions: Drug: High dose vehicle control

INTERVENTIONS:
Drug: Low dose ORTD-1 — Once weekly, single subcutaneous injection of ORTD-1 at a volume of 0.45 mL. Six weekly treatments; 28-day follow-up period.
  Other Names: ORTD-1
  Arms: ORTD-1-Low Dose
Drug: Low dose vehicle control — Once weekly subcutaneous injection of vehicle at a volume of 0.45 mL. Six weekly treatments; 28-day follow-up period.
  Other Names: Placebo
  Arms: Vehicle Control -Low Dose
Drug: High dose ORTD-1 — Two subcutaneous injections of ORTD-1 at two injection sites once weekly; 0.90 mL of ORTD-1 per each subcutaneous injection. Six weekly treatments; 28-day follow-up period.
  Other Names: ORTD-1
  Arms: ORTD 1-High Dose
Drug: High dose vehicle control — Two subcutaneous injections of vehicle at two injection sites once weekly; 0.90 mL of vehicle per each subcutaneous injection. Six weekly treatments; 28-day follow-up period.
  Other Names: Placebo
  Arms: Vehicle Control -High Dose

SUMMARY:
This is a randomized, vehicle controlled, double-blind, repeat dose comparative study in patients with rheumatoid arthritis (RA) under management with DMARDs and with persistent disease activity. The goal of this study is to evaluate the safety, tolerability and pharmacokinetics of 6 weekly repeat doses of ORTD-1.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age or older, males or females.
* Diagnosed rheumatoid arthritis per the American Rheumatism Association 1987 classification criteria of at least 6 months duration.
* Disease activity defined as:

  * erythrocyte sedimentation rate (ESR) > 24 mm or serum C-reactive protein level ≥ 1.2 times (X) the upper limit of normal (ULN), and
  * DAS28-CRP score ≥ 2.6 and < 5.1
* Current regimen of DMARDs that may include methotrexate, sulfasalazine, hydroxychloroquine, leflunomide and/or azathioprine, alone or in combination.
* No change in DMARD dose(s) within 4 weeks prior to Screening.
* May be receiving a stable regimen (of at least 4 weeks duration) of concomitant NSAIDs.
* Women of child-bearing potential (WOCBP), defined as a sexually mature woman not surgically sterilized, or not post-menopausal for at least 12 consecutive months. Female subjects must:

  * Not be lactating; not be pregnant upon enrollment.
  * Agree to use highly effective methods of birth control throughout the study. Highly effective methods of contraception include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation by oral, intravaginal, or transdermal administration; progestogen-only hormonal contraception associated with inhibition of ovulation by oral, injectable, or implantable administration; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; partner vasectomy; or total abstinence (only if total abstinence is an established method and lifestyle of the subject).
  * Patients already using hormonal contraception at the time of screening will be eligible but will not initiate hormonal contraception in order to participate in the study.
  * Agree to use highly effective methods of birth control for at least 6 months after the last dose of investigational product.
* Male subjects must refrain from donating sperm or fathering a child during the study.
* Male subjects must use barrier contraception throughout the course of the study.
* Signed and dated informed consent.

Exclusion Criteria:

* Prior therapy with any biologic therapeutic within 3 months prior to enrollment, or in the case of Rituxan (rituximab), this period must be at least 12 months.
* History of or current clinical fibromyalgia or Juvenile Idiopathic Arthritis (JIA).
* Positive diagnosis of SLE.
* Patients with Type 1 or Type 2 Diabetes Mellitus.
* Patients with psoriasis.
* Patients with skin condition(s) or visible abnormalities at or near potential sites of injection (right and left abdomen; right and left thigh) that could mask the assessment of safety.
* Acute illness including current or chronic infections requiring antibiotics, or symptoms of a resolving illness, within 2 weeks prior to study.
* Any investigational drug within 3 months prior to study.
* Patients may not be receiving systemic corticosteroid therapy with the exception of inhaled corticosteroids for the treatment of asthma.
* Any clinically relevant abnormality as assessed by the Investigator, on screening history, physical exam, clinical laboratory, chest X-ray, or ECG, other than values consistent with rheumatoid arthritis, with the exception that liver function tests (ALP, ALT, AST) may be up to 1.5 times (X) the upper limit of normal (ULN).
* Positive serological test for HCV, HBsAg, HBcAg, HIV.
* QuantiFERON-positive patients may be enrolled with documented evidence that they have completed a prescribed course of antituberculous therapy.
* History of cardiovascular disease with New York Heart Association (NYHA) functional class II or greater; or history of stroke, or uncontrolled hypertension.
* History of lymphoproliferative disease, or organ allograft.
* Pregnancy or lactation, or WOCBP not currently using contraceptives or male partners of WOCBP not currently using contraceptives.
* History of cancer (except for in situ cancer, or limited stage cancer of the cervix, head and neck (squamous cell), thyroid, or skin (non-melanomatous) curatively treated with no sign of disease for > 5 years).
* Any physical or psychological condition that might prevent complete participation in the study, in the view of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of ORTD-1 measured by the number of patients with adverse events | 10 weeks
  Safety will be assessed throughout the duration of the study (weeks 1 through 10) by monitoring of adverse events.

SECONDARY OUTCOMES:
Immunogenicity by measurement of anti-drug antibodies | Weeks 1, 3, 5, and 10
  Immunogenicity is the measurement of anti-drug (ORTD-1) antibodies (ADA) in serum. ADA samples will be analyzed from the change in baseline (Visit 1) using descriptive statistics (mean, median, range and standard deviation).
Serum concentration of ORTD-1 from baseline | 10 weeks
  Serum concentration will be measured from the change in baseline (Visit 1) using descriptive statistics (mean, median, range and standard deviation).
Cmax of ORTD-1 | Week 1 through week 6
  Cmax (maximum plasma concentration) will be measured using the arithmetic mean, standard deviation (SD), coefficient of variation (CV) (%), median, minimum, and maximum.
Tmax of ORTD-1 | Week 1 through week 6
  Tmax (time of maximum plasma concentration) will be measured using the arithmetic mean, standard deviation (SD), coefficient of variation (CV) (%), median, minimum, and maximum.

OTHER OUTCOMES:
Change from baseline in disease activity | Weeks 1, 3, 5, and 10
  Disease activity score with C-reactive protein (DAS28-CRP) and ESR (Erythrocyte sedimentation rate) will be evaluated from the change in baseline (Visit 1) to Visit 9 (last patient visit). 28 joints are evaluated in the DAS28-CRP (Proximal interphalangeal, metacarpophalangeal, wrists, elbows, shoulders, knees) for swelling and tenderness. The overall calculated value for DAS28-CRP uses the number of swollen and tender joints, the value recorded from the patient's CRP, and the Global Health patient assessment (0-100 mm; where 0 is very good and 100 is very bad health condition).

CONTACTS AND LOCATIONS:
Overall Officials: William Stohl, M.D., Ph.D., Principal Investigator — Keck School of Medicine of USC Division of Rheumatology
Locations (3):
- United States (3):
  - Keck School of Medicine of USC Division of Rheumatology, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - Advanced Pharma CR, LLC, Miami, Florida